CLINICAL TRIAL: NCT04537975
Title: A Randomized Clinical Trial of CLR2.0 Hemofiltration Treatment (C2Rx) in Severe or Critically Ill Adults With COVID-19 Infection
Brief Title: C2Rx Hemofiltration Treatment in Severe or Critically Ill Adults With COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn (Study was withdrawn by Sponsor because of change in regulatory strategy.)
Sponsor: SeaStar Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-01-004
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Continuous Renal Replacement Therapy; Pulmonary Edema; COVID-19
MeSH Terms: conditions — Pulmonary Edema; COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- C2Rx (Active Comparator): Hemofiltration device
  Interventions: Device: C2Rx
- Standard of Care (SOC) (Active Comparator): Standard of Care based on protocol inclusion/exclusion criteria
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: C2Rx — Hemofiltration
  Arms: C2Rx
Other: Standard of Care (SOC) — Standard of care that excludes any protocol restrictions.
  Arms: Standard of Care (SOC)

SUMMARY:
The clinical trial will evaluate the short term and extended impact on on respiration, pulmonary function and cardiovascular function in C2Rx treatment verse Standard of Care (SOC) in critically ill adults with COVID-19 infections .

ELIGIBILITY:
Inclusion Criteria:

* A patient, or legal authorized representative (LAR), has provided informed consent and a written informed consent form.
* Positive COVID-19 test.
* Must be receiving medical care in an intensive care nursing situation.
* Respiratory failure due to COVID-19 disease requiring invasive mechanical ventilation. This care may include but is not required to include the use of dexamethasone.
* Within 18 hours of tracheal intubation to support invasive mechanical ventilation. A goal of this study is that T0 will occur within 24 hours of tracheal intubation to support invasive mechanical ventilation.
* Age 18 to 80 years.
* Males and females (females of childbearing potential who are not pregnant confirmed by a negative serum pregnancy test) and not lactating if recently post-partum).
* Intent to deliver full supportive care through aggressive management utilizing all available therapies for a minimum of 96 hours.

Exclusion Criteria:

* Cardiovascular instability that precludes initiation of hemofiltration.
* Irreversible brain damage based on available historical and clinical information.
* Presence of any solid organ transplant at any time.
* Patients with stem cell transplant in the previous 100 days or who have not engrafted.
* Acute or chronic use of circulatory support device such as extracorporeal membrane oxygenation (ECMO), left ventricular assist devices (LVADs), right ventricular assist devices (RVADs), biventricular assist devices (BIVADs).
* Metastatic malignancy which is actively being treated or may be treated with chemotherapy or radiation during the subsequent three-month period after study treatment.
* Chronic immunosuppression defined as use of any immunosuppressant medications (cyclophosphamide, azathioprine, methotrexate, rituximab, mycophenolate, cyclosporine); prednisone use is excepted.
* Patient is moribund or chronically debilitated for whom full supportive care is not indicated.
* Concurrent enrollment in another interventional clinical trial except trials of COVID-19 convalescent plasma, anti-severe acute respiratory syndrome (SARS)-CoV2 monoclonal antibodies, or RemdesivirTM. Patients enrolled in observational studies (without the use of an investigative device or drug), are allowed to participate. Any communication between the Principal Investigator (PI) of this Protocol and the PI of any other clinical study will include the Medical Director of the Sponsor; all such correspondence will be documented.
* Any reason the Investigator deems exclusionary

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Oxygenation Function | Up to 72 hours
  Change in patient Arterial Oxygen Partial Pressure (PaO2)/Fractional Inspired Oxygen (FiO2) Ratio

SECONDARY OUTCOMES:
Pulmonary Compliance of Respiratory System (CRS) | Up to 96 hours
  Change in patient oxygenation
Survival | 30 days and 60 days
  Change in the total number of patients that survived
Hospital Costs 1 | Out to 60 days
  Change in Hospital Utilization of ventilators (days)
Cardiovascular Vasoactive-Inotropic Score (VIS) | Up to 96 hours
  Change in score based on the calculation of the following medications used: dopamine dose (µg/kg/min) + dobutamine dose (µg/kg/min) + 100 x adrenaline dose (µg/kg/min) + 100 x noradrenaline dose (µg/kg/min) + 10 x milrinone dose (µg/kg/min) + 10.000 x vasopressin dose (U/kg/min)
Hospital Costs 2 | Out to 60 days
  Change in Hospital Utilization of vasopressor medication (days without use)
Hospital Costs 3 | Out to 60 days
  Change in Hospital Utilization of Intensive Care Unit (ICU) Hospital free days
Hospital Costs 4 | Out to 60 days
  Change in Hospital Utilization of Renal Replacement Therapy (days on therapy)
Hospital Costs 5 | Out to 60 days
  Change in Hospital Utilization (days hospitalized)

OTHER OUTCOMES:
Inflammatory mediators in blood | Out to 14 hours
  Changes in inflammatory mediators detected by Immunoassay of Multianalyte Panel - MAP Laboratory Panel of 253 analytes.
Cytokine Sieving Effects | Out to 8 hours
  Change in cytokine levels obtained from plasma and blood collected prior to and after filter. Analyte concentrations in ultrafiltrate and plasma, expressed in the same concentration units, will be aggregated as a ratio of ultrafiltrate concentration to plasma concentration to yield a unitless Sieving Coefficient (SC). SC is an index of membrane function.
Specific Blood Indicators 1 | Out to 14 hours
  Change in blood Ferritin (mg/mL)
Specific Blood Indicators 2 | Out to 14 hours
  Change in blood Interleukin-6 (pg/mL)
Specific Blood Indicators 3 | Out to 14 hours
  Change in blood C-reactive protein (CRP) (mg/L)
Specific Blood Indicators 4 | Out to 14 hours
  Change in blood Lactate Dehydrogenase (LDH) (U/L)
Specific Blood Indicators 5 | Out to 14 hours
  Change in blood D-dimer (mcg/L*FEU2)
Specific Blood Indicators 6 | Out to 14 hours
  Change in blood White Blood Cell (WBC) count (%)
Specific Blood Indicators 7 | Out to 14 hours
  Change in blood Neutrophil count (%)
Specific Blood Indicators 8 | Out to 14 hours
  Change in blood lymphocyte count (%).
Hospital Acquired Infections (HAI) /Sepsis | 30 and 60 days
  Change in the duration of days of diagnosed HAI/ Sepsis infections
Composite Recovery | Up to 30 days
  Duration without Respiratory Replacement Therapy (RRT), ventilator, and time to discharge
Composite Survival | 30 and 60 days
  Survival without Respiratory Replacement Therapy (RRT), ventilator, or time to Long Term Care (LTC)
Composite Non-Recovery | Up to 60 days
  Survival with Respiratory Replacement Therapy (RRT), ventilator or in Long Term Care (LTC)

IPD SHARING:
Plan to Share IPD: No